CLINICAL TRIAL: NCT05260333
Title: Use of a Pocket-device Point-of-care Ultrasound to Assess Cervical Dilation in Labor: Correlation and Patient Experience
Brief Title: Sound Check-Correlation Between Transperineal and Digital Cervical Exam in 3rd Trimester Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Leah Antoniewicz, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: H-50937
Record Dates: First submitted 2022-02-16; First posted 2022-03-02 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cervix; Pregnancy
Keywords: transperineal; ultrasound; cervix; labor

STUDY DESIGN:
Intervention Model Description: Patients will have a transperineal ultrasound followed by a traditional digital cervical exam.
Masking Description: The investigator will not know the digital cervical exam value.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transperineal ultrasound cervical exam followed by Digital (manual) cervical exam (Experimental): Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound. Patients will then undergo traditional digital cervical exam via examiner's fingers.
  Interventions: Device: Butterfly iQ transperineal ultrasound exam

INTERVENTIONS:
Device: Butterfly iQ transperineal ultrasound exam — Transperineal ultrasound

SUMMARY:
The primary purpose of this study is to compare the accuracy of the Butterfly iQ pocket ultrasound with the digital cervical examination in the third trimester cervix. The secondary aim of this study is to compare discomfort or the two cervical exam methods and determine if patients have a preference for one over the other.

DETAILED DESCRIPTION:
Patients in the 3rd trimester that require a digital cervical exam (DCE) for assessment of labor will be approached. After informed consent is obtained, one of two study investigators will perform a transperineal ultrasound (TPUS) using the glove-covered Butterfly iQ+ probe. The Butterfly iQ+ does not have a transperineal probe or setting, therefore, the "bladder" preset setting will be used. The "bladder" setting has been predetermined to provide the best cervical images. This pocket ultrasound is FDA-approved and is the standard of care for point of care ultrasounds in many institutions and is already used in our department. The TPUS will be performed by 1 of the 2 investigators with digital calipers. There will be 3 measurements: dilation, effacement, and station. The dilation measurements with be made from the inside margins of the cervix . Effacement will be measured by marking the thinnest and most easily imaged lip of the cervix. Zero station will be assumed to be 5 cm above the perineum, with distances from 6-10 cm corresponding to -1 to -5 station clinically. An independent, blinded examiner will then perform a traditional digital cervical exam, which will be recorded in EPIC. The study investigators will be blinded to the DCE measurement until the end of the study. The patient will act as their own control. Additionally, the investigators will collect EGA, race, ethnicity, age, BMI, and indication for assessment of the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester presenting for assessment of labor or admitted for labor and delivery.

Exclusion Criteria:

* Second trimester (less than 28 weeks)
* BMI>50
* Does not wish to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah W Antoniewicz, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richey SD, Ramin KD, Roberts SW, Ramin SM, Cox SM, Twickler DM. The correlation between transperineal sonography and digital examination in the evaluation of the third-trimester cervix. Obstet Gynecol. 1995 May;85(5 Pt 1):745-8. doi: 10.1016/0029-7844(95)00027-o. PMID 7724106
- [Background] Mahony BS, Nyberg DA, Luthy DA, Hirsch JH, Hickok DE, Petty CN. Translabial ultrasound of the third-trimester uterine cervix. Correlation with digital examination. J Ultrasound Med. 1990 Dec;9(12):717-23. doi: 10.7863/jum.1990.9.12.717. PMID 2277401
- [Background] Newton ER. Chorioamnionitis and intraamniotic infection. Clin Obstet Gynecol. 1993 Dec;36(4):795-808. doi: 10.1097/00003081-199312000-00004. PMID 8293582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled in April of 2022, and last patient was seen in July of 2022.
Groups:
- Transperineal Ultrasound and Digital Cervical Exam: Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound followed by a traditional digital cervical exam.
  Butterfly iQ transperineal ultrasound exam: Transperineal ultrasound
Period: Overall Study
Arm/Group | Transperineal Ultrasound and Digital Cervical Exam
Started (The patients acted as there own control. 30 patients were enrolled, but a total of 60 exams (1 TPUS and 1 SVE) were performed.) | 30
Transperineal Ultrasound (The patients acted as there own control. 30 patients were enrolled, but a total of 60 exams (1 TPUS and 1 SVE) were performed.) | 30
Digital Cervical Exam (The patients acted as there own control. 30 patients were enrolled, but a total of 60 exams (1 TPUS and 1 SVE) were performed.) | 30
Completed (The patients acted as there own control. 30 patients were enrolled, but a total of 60 exams (1 TPUS and 1 SVE) were performed.) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Transperineal Ultrasound Cervical Exam and Digital (Manual) Cervical Exam: Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound and then undergo traditional digital cervical exam via examiner's fingers..
  Butterfly iQ transperineal ultrasound exam: Transperineal ultrasound
Arm/Group | Transperineal Ultrasound Cervical Exam and Digital (Manual) Cervical Exam
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants] — Collected from chart
  Participants
    <=18 years | 0
    Between 18 and 65 years | 30
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Cervical Dilation [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Cervical Dilation Via Butterfly iQ Pocket Ultrasound in Centimeters
Description: Dilation was measured on the day of the exam in centimeters. A correlation coefficient was then calculated to determine the relationship between the two exams.
Time Frame: 1 day
Population: The patients served as their own control.
Measure: Median (Full Range); unit: centimeters
Groups:
- Transperineal Ultrasound Cervical Exam Dilation; Digital (Manual) Cervical Exam Dilation: Diameter of cervix in centimeters
Arm/Group | Transperineal Ultrasound Cervical Exam Dilation | Digital (Manual) Cervical Exam Dilation
Number analyzed (Participants) | 30 | 30
centimeters | 5.1 [0 to 10] | 5 [0 to 10]
Statistical Analysis 1: Comparison: Transperineal Ultrasound Cervical Exam Dilation; Test type: Other; p = .0001, Wilcoxon (Mann-Whitney); correlation coefficient = 0.81

2. Secondary Outcome: Discomfort Scale
Description: 3-point Likert scale (0 = no discomfort, 3 = maximum) discomfort on questionnaire.
Time Frame: 1 day
Measure: Median (Full Range); unit: score on a scale
Groups:
- Transperineal Ultrasound Cervical Exam Followed by Digital (Manual): Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound. Then patients will undergo traditional digital cervical exam via examiner's fingers.
Arm/Group | Transperineal Ultrasound Cervical Exam Followed by Digital (Manual)
Number analyzed (Participants) | 30
score on a scale
  Transperineal | 0 [0 to 2]
  Digital | 2 [0 to 2]

3. Secondary Outcome: Preference for 1 Exam Over the Other
Description: Patients were asked if they had a preference and circled yes or no on questionnaire
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Transperineal Ultrasound Cervical Exam Followed by Digital (Manual): Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound followed by digital cervical exam.
Arm/Group | Transperineal Ultrasound Cervical Exam Followed by Digital (Manual)
Number analyzed (Participants) | 30
Participants
  Preferred TPUS | 30
  Preferred Digital | 0

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Transperineal Ultrasound Cervical Exam: Patients will undergo transperineal cervical exam via Butterfly iQ ultrasound.
  Butterfly iQ transperineal ultrasound exam: Transperineal ultrasound
- Digital (Manual) Cervical Exam: Patients will undergo traditional digital cervical exam via examiner's fingers.
  Butterfly iQ transperineal ultrasound exam: Transperineal ultrasound
Arm/Group | Transperineal Ultrasound Cervical Exam | Digital (Manual) Cervical Exam
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT05260333/Prot_SAP_001.pdf